CLINICAL TRIAL: NCT06339216
Title: A Phase II Clinical Study of Adebrelimab Injection in Combination With Apatinib and Paclitaxel for Injection (Albumin-bound) as Second-line Therapy in Patients With Advanced Gastric Cancer Who Had Previously Received Immunotherapy.
Brief Title: A Clinical Study of Adebrelimab Combined With Apatinib and Paclitaxel in Patients With Advanced Gastric Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-GC-II-011
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: Second-line treatment population,Patients who have received immunotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab+Apatinib+Paclitaxel for Injection(Albumin Bound) (Experimental): Adebrelimab injection was started on Day 1 of each cycle, followed 30 minutes later by intravenous drip of Paclitaxel for Injection(Albumin Bound). Combined treatment for 6 to 8 weeks, after efficacy evaluation, the investigator decides the subsequent treatment regimen, or until disease progression, toxicity intolerance, initiation of new anti-tumor therapy, withdrawal of informed consent, or the investigator judges that the subject needs to withdraw from the study treatment. Following RECISTv1.1 defined progression (as assessed by the investigator), study drug may continue if the investigator assesses that the subject is still receiving clinical benefit and tolerates study treatment.
  Interventions: Drug: Adebrelimab+Apatinib+Paclitaxel for Injection(Albumin Bound)

INTERVENTIONS:
Drug: Adebrelimab+Apatinib+Paclitaxel for Injection(Albumin Bound) — Adebrelimab injection：Intravenous infusion, fixed dose 1200 mg, Day 1, Q3W. Until disease progression or intolerable toxicity occurs, the infusion should be administered over 30 to 60 minutes and over a maximum of 2 hours. When adalimumab is administered in combination with chemotherapy, Adebrelimab should be administered as an intravenous infusion first, followed by chemotherapy at least 30 minutes apart.
  Apatinib mesylate：Administered orally, 250 mg/time, once daily, orally, half an hour after meals (the time of daily administration should be as same as possible), with warm boiled water, the missed dose of Apatinib during the course of treatment cannot be supplemented.
  Paclitaxel for Injection(Albumin Bound)：Intravenous infusion, 250 mg/m2, day 1, Q3W, intravenous drip over 30 minutes.

SUMMARY:
Phase II Clinical Study of Adebrelimab Combined with Apatinib and Paclitaxel for Injection(Albumin Bound) as Second-line Therapy in Patients with Advanced Gastric Cancer Previously Treated with Immunotherapy

DETAILED DESCRIPTION:
To observe and evaluate the efficacy of Adebrelimab combined with Apatinib and Paclitaxel for Injection(Albumin Bound) in second-line treatment of advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18 years and older, male or female.
2. patients with pathologically or cytologically confirmed gastric cancer (GC) or gastroesophageal junction cancer (GEJ).
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
4. measurable lesions that meet RECIST1.1 criteria.
5. Patients with gastric cancer who have progressed on first-line immunotherapy have achieved CR or PR or SD ≥ 3 months on the first immunotherapy;
6. expected survival ≥ 3 months;
7. Normal function of major organs, no severe blood, heart, lung, liver and kidney dysfunction and immunodeficiency diseases. Laboratory tests were to meet the following requirements: neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109/L) (no growth factors used within 14 days); platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L) (no corrective treatment used within 7 days); hemoglobin (Hb) ≥ 9 g/dL (90 g/L) (no corrective treatment used within 7 days); serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min; total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN); aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) levels ≤ 2.5 times the upper limit of normal (ULN), and ≤ 5 × ULN for patients with liver metastases. Serum Cr ≤ 1.5 times ULN, endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula); Normal urine routine, or urine protein < (+ +), or 24-hour urine protein < 1.0g;
8. normal coagulation function, no active bleeding and thrombosis disease: international normalized ratio INR ≤ 1.5 × ULN; partial thromboplastin time APTT ≤ 1.5 × ULN; prothrombin time PT ≤ 1.5ULN;
9. Patients with potential fertility need to use a medically recognized contraceptive (such as intrauterine device, contraceptives or condoms) during study treatment and within 3 months after the end of study treatment; and must have a negative serum HCG test within 72 hours before study enrollment; and must be non-lactating. I agree and have signed an informed consent form and am willing and able to comply with scheduled visits, study treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. history of gastrointestinal perforation and/or fistula within 6 months before the first dose;
2. presence of uncontrollable pleural effusion, pericardial effusion, or abdominal effusion requiring repeated drainage;
3. previous history of hypersensitivity to monoclonal antibodies, any component of adalimumab, and nab-paclitaxel;
4. received any of the following treatments: a. previously received immunotherapy with serious adverse reactions; b. received any investigational drug within 4 weeks before the first use of study drug; c. enrolled in another clinical study at the same time, unless it was an observational (non-interventional) clinical study or interventional clinical study follow-up; d. received the last dose of anticancer therapy ≤ 3 weeks before the first use of study drug and received fixed-field palliative radiotherapy ≤ 2 weeks before the first study intervention treatment; e. subjects who required corticosteroids (> 10 mg prednisone equivalent dose per day) within 2 weeks before the first use of study drug. Other special situations require communication with the sponsor. In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticotropic hormone replacement at doses > 10 mg/day prednisone efficacy dose are allowed; f. those who have received anti-tumor vaccines or live vaccines within 4 weeks before the first dose of study drug; g. major surgery or severe trauma within 4 weeks before the first dose of study drug;
5. previous anti-tumor treatment toxicity did not recover to ≤ CTCAE grade 1 (except alopecia) or the level specified in the inclusion/exclusion criteria;
6. patients with central nervous system metastases;
7. History of active autoimmune diseases, autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes): except leukoplakia or recovered childhood asthma/allergy, patients who do not require any intervention after adulthood: autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; type I diabetes treated with stable doses of membrane insulin;
8. history of immunodeficiency, including HIV test positive, or suffering from other acquired, congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation;
9. the subject has cardiovascular clinical symptoms or diseases that are not well controlled, including but not limited to: (1) heart failure above NYHA II; (2) unstable angina pectoris; (3) myocardial infarction within 1 year; (4) clinically significant supraventricular or ventricular arrhythmia that remains poorly controlled without or after clinical intervention;
10. Urine routine showed urine protein ≥ + + and confirmed 24-hour urine protein > 1.0g;
11. Patients with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds), bleeding tendency or receiving thrombolytic or anticoagulant therapy are allowed to receive low-dose low-molecular-weight heparin or oral aspirin to prevent anticoagulant therapy during the trial;
12. Patients who have experienced clinically significant bleeding symptoms or definite bleeding tendency within 3 months before randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or suffering from vasculitis, etc. If fecal occult blood is positive at baseline, they can be reexamined. If it is still positive after reexamination, gastroscopy should be performed when necessary in combination with clinical judgment;
13. Accompanied by active ulcers, unhealed wounds or fractures;
14. Patients with hypertension, and can not be well controlled by antihypertensive drug treatment (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
15. serious infection (CTCAE > 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging showed active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first use of the study drug or the need for oral or intravenous antibiotic treatment, except for the prophylactic use of antibiotics;
16. Patients with a history of interstitial lung disease (except radiation pneumonitis and non-infectious pneumonitis who have not used hormone therapy);
17. Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than 1 year ago but without regular treatment;
18. Patients who have been diagnosed with any other malignant tumor within 5 years before the first use of the study drug, except for malignant tumors with low risk of metastasis and death (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ;
19. Pregnant or lactating women;
20. The investigator judges that the subject has other factors that may cause the subject to be forced to terminate the study halfway, such as having other serious diseases (including mental illness) requiring concomitant treatment, severely abnormal laboratory values, family or social factors, which may affect the subject 's safety or the collection of trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 3 years
  The proportion of patients with a confirmed complete response or partial response

SECONDARY OUTCOMES:
PFS | up to 3 years
  The time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first
DCR | up to 3 years
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease
OS | up to 3 years
  The time from randomization to death from any reason

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, Doctor, Study Chair — Chinese PLA General Hospital